CLINICAL TRIAL: NCT06843668
Title: Efficacy and Safety of Different Dosing Strategies of Colistin in Multidrug-Resistant Gram-Negative Bacilli Infections in Critically Ill Patients
Brief Title: Different Dosing Strategies of Colistin in Multidrug-Resistant Gram-Negative Bacilli Infections
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mona Mohammed El-Tamalawy, Lecturer of Clinical Pharmacy, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-04-Q001
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-02

CONDITIONS: Critical Ill Patients; Multi Drug Resistant

STUDY DESIGN:
Intervention Model Description: This is a prospective, single blind, randomized, comparative intervention study .
Who Masked: Participant
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The EMA (fixed dose) colistin group (Experimental): The EMA colistin group will receive I.V colistin using fixed dose strategy.
  Interventions: Drug: EMA colistin dosing strategy
- US FDA (weight-based dose) colistin group (Active Comparator): The weight-based colistin group will receive I.V. colistin using weight based dosing strategy.
  Interventions: Drug: US FDA colistin dosing strategy

INTERVENTIONS:
Drug: EMA colistin dosing strategy — The EMA colistin group will receive I.V colistin based on creatinine clearance (mL/min) level , with fixed loading dose 9 MIU equivalent to 300 mg of colistin-based activity (CBA). The maintenance dose will be administered after 12 h following the loading dose over 1 h every 12h (twice daily).
  Arms: The EMA (fixed dose) colistin group
Drug: US FDA colistin dosing strategy — The weight-based colistin group will receive I.V. colistin based on the lower (ideal body weight or actual body weight) with a loading dose of (4) X (patient weight in kg). Loading dose might exceed 300 mg.
  Arms: US FDA (weight-based dose) colistin group

SUMMARY:
Nosocomial infections caused by multi-drug-resistant (MDR) and extensively drug-resistant (XDR) Gram-negative pathogens represent a major threat worldwide. The increasing trend of multi-drug resistance in Gram-negative bacteria (MDR-GNB) poses a particularly acute challenge to health systems especially in critically ill patients.

Patients in intensive care units (ICUs) have encountered an increasing emergence and spread of antibiotic-resistant pathogens. In Saudi Arabia mainly MDR-GNB such as Acinetobacter Baumannii, Pseudomonas Aeruginosa, Klebsiella Pnemoniae and Enterobacter are observed in ICUs.

Polymyxins are the last line therapy in the treatment of infection caused by these MDR-GNB. Colistin is the most widely used polymyxin antibiotic, it is administered as inactive prodrug colistimethate sodium (CMS) that is hydrolyzed to an active moiety of colistin base activity (CBA). It acts as cationic detergent and damages bacterial cytoplasmic membrane causing leaking of intracellular substances and then cell death.

During the first years of their use, polymyxin-associated neurotoxicity occurred in patients with an incidence as high as 27% following parenteral administration. However, other retrospective clinical trials have not exposed neurotoxicity to be a major concern. On the other hand, nephrotoxicity is by far the most common and dose-limiting side effect associated with parenteral polymyxins, with incidence rates in patients as high as 60%. Despite the high incidence of colistin induced nephrotoxicity, in 2012, the World Health Organization (WHO) reclassified polymyxins as critically important for the management of MDR-GNB infection, renewing the interest in these antibiotics.

To the best of our knowledge no study compared the efficacy and safety of both dosing strategies in critically ill patients. Moreover, there is still a lack of evidence on the efficacy and safety of both dosing strategies in obese patients. Therefore, this study aims at comparing the efficacy and toxicity of both strategies in colistin dosing (the fixed dose and the weight-based dosing) in obese patients and non- obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years old.
* Patients who will be treated with CMS for MR GNB infections.
* Patients who are admitted to the ICUs.

Exclusion Criteria:

* Known hypersensitivity to colistin.
* Pregnant and lactating women.
* Patients who are treated with colistin for < 24 hours.
* Patients with myasthenia gravis or concomitant anesthetics or neuromuscular blocking drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Clinical and microbiological success in eradication of infection reported as the number and percentage of patients with successful clinical improvement and microbiological clearance (Efficacy). | 14 days post colistin initiation.
  having a white blood cell count (WBC) of less than 12,000 cells/mm3 or a ≥ 25% reduction in WBC, being afebrile for ≥ 48 h,.
  • Microbiological clearance will be defined as eradication of the original causative organism from subsequent blood cultures by day 14 of therapy.

SECONDARY OUTCOMES:
Nephrotoxicity (Safety) | 14 days
  nephrotoxicity was defined as doubling of baseline serum creatinine level or drop-in baseline creatinine clearance rate by ≥50%.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Shams, Professor, Principal Investigator — Mansoura University
Locations (1):
- King Fahad Specialist Hospital, Buraidah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Nation RL, Turnidge JD, Milne RW, Coulthard K, Rayner CR, Paterson DL. Colistin: the re-emerging antibiotic for multidrug-resistant Gram-negative bacterial infections. Lancet Infect Dis. 2006 Sep;6(9):589-601. doi: 10.1016/S1473-3099(06)70580-1. PMID 16931410
- [Background] Maraki S, Mantadakis E, Nioti E, Samonis G. Susceptibility of 2,252 Pseudomonas aeruginosa Clinical Isolates Over 4 Years to 9 Antimicrobials in a Tertiary Greek Hospital. Chemotherapy. 2014;60(5-6):334-41. doi: 10.1159/000437252. Epub 2015 Aug 18. PMID 26302835